CLINICAL TRIAL: NCT05763667
Title: A Randomized, Controlled, Observer-blinded Pilot Trial of Laparoscopic Large Volume, Multisite Transversus Abdominal Plane (TAP) Block With Liposomal Bupivacaine in Patients Undergoing Minimally Invasive Hysterectomy for Endometrial Cancer
Brief Title: Pilot: Intraoperative TAP Block and Post-operative Pain Control for Minimally Invasive Hysterectomy for Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Pain; Gynecologic Cancer
Keywords: hysterectomy; minimally invasive surgery; TAP block; endometrial cancer; endometrial intraepithelial neoplasia
MeSH Terms: conditions — Pain, Postoperative; Endometrial Neoplasms; Endometrial Hyperplasia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Potential subjects will be identified in the GYN specialty clinics at Tufts Medical Center and approached for possible study participation. Eligibility criteria will be assessed by the PI or co-I. Eligible subjects who wish to participate in the study will be consented for the study by the PI or co-I. Informed consent for the study may be obtained up to the day of the surgery, prior to anesthesia induction. The following demographics will be collected from the medical record and de-identified: age, race, ethnicity, height, weight, ASA class.
  On the day of surgery, the subject will be randomized using a random number generator to one of 3 groups:
  1. No TAP block
  2. TAP block with liposomal and plain bupivacaine: 20 mL liposomal bupivacaine, 30 mL 0.25% bupivacaine, 150 mL normal saline (200 mL total)
  3. TAP block with plain bupivacaine alone: 60 mL of 0.25% bupivacaine, 140 mL of normal saline (200 mL total)
Who Masked: Participant, Outcomes Assessor
Masking Description: The pharmacy will prepare the solutions for groups 2 and 3, reflecting the usual practice of this PI and his mentees. No solution will be prepared for group 1, as this is a form of standard care for patients undergoing minimally invasive hysterectomy. As the liposomal bupivacaine has a cloudy appearance whereas plain bupivacaine and saline are clear, the surgeon will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- No TAP block (No Intervention)
- TAP block with liposomal and plain bupivacaine (Active Comparator)
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacain
- TAP block with plain bupivacaine alone (Active Comparator)
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal bupivacaine is FDA-approved for use single-dose infiltration in adults to produce postsurgical local analgesia and as an interscalene brachial plexus nerve block to produce postsurgical regional analgesia.
  The solution will be placed into 20 mL syringes on 18-gauge needles for injection. The injections will be performed percutaneously by the surgeon along the midaxillary line at 4 equidistant points from the anterior superior iliac spine to the costal margin, as well as a single injection subcostally at the anterior axillary line. 20 mL will be injected at each site, 5 sites per side bilaterally, total of 10 sites. The depth of injection will be judged by laparoscopic visualization of a diffuse bulge during injection, indicating injection in the correct plane, just superficial to the transversus abdominis muscle.
  Other Names: Exparel
  Arms: TAP block with liposomal and plain bupivacaine
Drug: Bupivacain — Bupivacaine is FDA-approved for use as a local or regional anesthetic for surgery. It is widely used in TAP blocks.
  The solution will be placed into 20 mL syringes on 18-gauge needles for injection. The injections will be performed percutaneously by the surgeon along the midaxillary line at 4 equidistant points from the anterior superior iliac spine to the costal margin, as well as a single injection subcostally at the anterior axillary line. 20 mL will be injected at each site, 5 sites per side bilaterally, total of 10 sites. The depth of injection will be judged by laparoscopic visualization of a diffuse bulge during injection, indicating injection in the correct plane, just superficial to the transversus abdominis muscle.
  Other Names: Bupivacaine
  Arms: TAP block with liposomal and plain bupivacaine; TAP block with plain bupivacaine alone

SUMMARY:
Modern postoperative pain management aims to optimizing pain relief while minimizing opiate usage. While opiates are effective for pain relief, they result in common adverse effects such as nausea, constipation, and urinary retention, and most importantly present a long-term risk of abuse and dependency. Commonly used approaches include non-opiate pain medications such as acetominophen and non-steroidal anti-inflammatory agents, as well as regional nerve blocks such as epidurals.

The transversus abdominis plane (TAP) block is a fascial plane block performed by injecting local anesthetic into the plane superficial to the transversus abdominis muscle where the anterior rami of the spinal nerves course to provide sensory innervation to the abdominal wall. The injections are generally placed either subcostally or at the midaxillary line bilaterally. The TAP block has been shown to be effective in reducing pain scores and opiate usage in some randomized studies but not others in patients undergoing various abdominal surgeries. There is great variation in method of administration, sites injected, and local anesthetics used, which may in part account for the heterogeneity of trial results.

DETAILED DESCRIPTION:
The investigators believe that the disappointing results thus far with TAP blocks in minimally invasive hysterectomy may relate to several factors. A combination of short and long-acting anesthetic agents may provide the optimal analgesic effect. Large volumes of injection may promote spread of the anesthetics for better coverage, especially as long-acting agents are known to diffuse minimally. Lastly, multiple injections may provide better coverage of the nerves that innervate the abdominal wall.

The investigators also believe that laparoscopic TAP blocks, administered by the surgeon, have advantages over the more commonly used ultrasound-guided approach typically performed by anesthesiologists. The laparoscopic approach is quick, on the order of a few minutes, whereas the ultrasound approach can be time-consuming. There is also less risk of visceral injury since the injection is performed under direct laparoscopic view. There are now 2 randomized studies suggesting that the laparoscopic approach is equivalent to the ultrasound approach.

An additional potential reason why most studies have been negative is that patients undergoing minimally invasive hysterectomy do not generally experience severe pain, making it more difficult to demonstrate pain reduction with any given intervention. However, the studies to date do indicate that these patients experience moderate pain and do use opiates. An intervention that markedly reduces or even eliminates opiate use would be of potential benefit.

The investigators have used a TAP block technique that is performed intraoperatively by the surgeon under direct laparoscopic view. The investigators use a mixture of plain and liposomal bupivacaine injected at multiple sites and in large volume to distribute the drugs widely, potentially resulting in longer and improved efficacy. This method has not been previously studied in a randomized trial. The investigators propose to demonstrate that this technique markedly decreases opiate usage and pain scores in patients undergoing minimally invasive hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. Patients undergoing laparoscopic or robotic hysterectomy; may include other procedures (e.g. lymph node removal)
3. Endometrial cancer or endometrial intraepithelial neoplasia
4. Able to consent to study

Exclusion Criteria:

1. Known clinically significant allergy to bupivacaine or liposomal bupivacaine
2. ASA IV or V
3. Emergency surgery
4. Current chronic opiate use
5. Current pregnancy or breastfeeding
6. Severe hepatic or renal impairment
7. Hysterectomy is not for endometrial cancer or endometrial intraepithelial neoplasia

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Reduced opiate use in both TAP block arms. | 7 days
  Demonstrate a statistically significant change in postoperative opiate use as measured in oral morphine milligram equivalents on postoperative days 0-7.

SECONDARY OUTCOMES:
Increase in opiate-free participants by day 7 | 7 days
  Demonstrate a change in proportion of subjects that are opiate-free on postoperative days 0-7.
Reduction in post-operative resting pain scores | 7 days
  Demonstrate a statistically significant change in maximum resting numeric rating scale (NRS) at the following time points in postoperative days: 0-1, 1-2, 2-3, 0-7.
Improvement in patient satisfaction regarding pain control | 7 days
  Demonstrate change in patient satisfaction with regard to pain control (very satisfied, satisfied, unsatisfied).
Incidence of Treatment-Emergent Adverse Events | 7 days
  Specific AEs measured will be nausea, headache, rash, itching, hematoma, ecchymosis, seizures

CONTACTS AND LOCATIONS:
Overall Officials: Young B Kim, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohel G, Kisselevitz R, Margalioth EJ, Schenker JG. Ascorbate-dependent lipid peroxidation in the human placenta and fetal membranes. Gynecol Obstet Invest. 1985;19(2):73-7. doi: 10.1159/000299011. PMID 3921439
- [Background] Cserhati G, Szilagyi J, Pongracz S. [Yersinia pseudotuberculosis infection]. Orv Hetil. 1982 Jun 6;123(23):1431-2. No abstract available. Hungarian. PMID 7050825
- [Background] Babazade R, Saasouh W, Naylor AJ, Makarova N, Udeh CI, Turan A, Udeh BL. The cost-effectiveness of epidural, patient-controlled intravenous opioid analgesia, or transversus abdominis plane infiltration with liposomal bupivacaine for postoperative pain management. J Clin Anesth. 2019 Mar;53:56-63. doi: 10.1016/j.jclinane.2018.10.003. Epub 2018 Oct 13. PMID 30326379
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Seitz F. Science, the universities, and society. Am Sci. 1968 Autumn;56(3):288-97. No abstract available. PMID 5684553
- [Background] Baeriswyl M, Kirkham KR, Kern C, Albrecht E. The Analgesic Efficacy of Ultrasound-Guided Transversus Abdominis Plane Block in Adult Patients: A Meta-Analysis. Anesth Analg. 2015 Dec;121(6):1640-54. doi: 10.1213/ANE.0000000000000967. PMID 26397443
- [Background] Ilfeld BM, Viscusi ER, Hadzic A, Minkowitz HS, Morren MD, Lookabaugh J, Joshi GP. Safety and Side Effect Profile of Liposome Bupivacaine (Exparel) in Peripheral Nerve Blocks. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):572-82. doi: 10.1097/AAP.0000000000000283. PMID 26204387
- [Background] Hamilton TW, Athanassoglou V, Trivella M, Strickland LH, Mellon S, Murray D, Pandit HG. Liposomal bupivacaine peripheral nerve block for the management of postoperative pain. Cochrane Database Syst Rev. 2016 Aug 25;2016(8):CD011476. doi: 10.1002/14651858.CD011476.pub2. PMID 27558150
- [Background] Ji YD, Harris JA, Gibson LE, McKinley SK, Phitayakorn R. The Efficacy of Liposomal Bupivacaine for Opioid and Pain Reduction: A Systematic Review of Randomized Clinical Trials. J Surg Res. 2021 Aug;264:510-533. doi: 10.1016/j.jss.2021.02.024. Epub 2021 Apr 13. PMID 33862580
- [Background] Wong KA, Cabrera AG, Argiroff AL, Pechman DM, Parides MK, Vazzana JT, Moran-Atkin EM, Choi JJ, Camacho DR. Transversus abdominis plane block with liposomal bupivacaine and its effect on opiate use after weight loss surgery: a randomized controlled trial. Surg Obes Relat Dis. 2020 Jul;16(7):886-893. doi: 10.1016/j.soard.2020.03.031. Epub 2020 Apr 10. PMID 32402732
- [Background] Truong A, Fleshner PR, Mirocha JM, Tran HP, Shane R, Zaghiyan KN. A Prospective Randomized Trial of Surgeon-Administered Intraoperative Transversus Abdominis Plane Block With Bupivacaine Against Liposomal Bupivacaine: The TINGLE Trial. Dis Colon Rectum. 2021 Jul 1;64(7):888-898. doi: 10.1097/DCR.0000000000002008. PMID 34086002
- [Background] Okamoto Y, Ota K. [Changes in calcium regulating hormone in osteoporosis]. Nihon Rinsho. 1994 Sep;52(9):2295-300. Japanese. PMID 7967071
- [Background] Fidkowski CW, Choksi N, Alsaden MR. A randomized-controlled trial comparing liposomal bupivacaine, plain bupivacaine, and the mixture of liposomal bupivacaine and plain bupivacaine in transversus abdominus plane block for postoperative analgesia for open abdominal hysterectomies. Can J Anaesth. 2021 Jun;68(6):773-781. doi: 10.1007/s12630-020-01911-1. Epub 2021 Jan 11. PMID 33432496
- [Background] Hutchins J, Delaney D, Vogel RI, Ghebre RG, Downs LS Jr, Carson L, Mullany S, Teoh D, Geller MA. Ultrasound guided subcostal transversus abdominis plane (TAP) infiltration with liposomal bupivacaine for patients undergoing robotic assisted hysterectomy: A prospective randomized controlled study. Gynecol Oncol. 2015 Sep;138(3):609-13. doi: 10.1016/j.ygyno.2015.06.008. Epub 2015 Jun 6. PMID 26056753
- [Background] Ghisi D, Fanelli A, Vianello F, Gardini M, Mensi G, La Colla L, Danelli G. Transversus Abdominis Plane Block for Postoperative Analgesia in Patients Undergoing Total Laparoscopic Hysterectomy: A Randomized, Controlled, Observer-Blinded Trial. Anesth Analg. 2016 Aug;123(2):488-92. doi: 10.1213/ANE.0000000000001267. PMID 27074894
- [Background] Kane SM, Garcia-Tomas V, Alejandro-Rodriguez M, Astley B, Pollard RR. Randomized trial of transversus abdominis plane block at total laparoscopic hysterectomy: effect of regional analgesia on quality of recovery. Am J Obstet Gynecol. 2012 Nov;207(5):419.e1-5. doi: 10.1016/j.ajog.2012.06.052. Epub 2012 Jun 29. PMID 22840413
- [Background] Bringer J, Klawatsch D, Jaffiol C, Orsetti A, Robin M, Mirouze J. [Comparison of various treatments for tumoral acromegaly. Study of initial prognostic factors]. Ann Endocrinol (Paris). 1983 Mar-Apr;44(2):107-14. No abstract available. French. PMID 6614855
- [Background] Calle GA, Lopez CC, Sanchez E, De Los Rios JF, Vasquez EM, Serna E, Arango AM, Castaneda JD, Vasquez RA, Gonzalez A, Escobar A, Almanza LA. Transversus abdominis plane block after ambulatory total laparoscopic hysterectomy: randomized controlled trial. Acta Obstet Gynecol Scand. 2014 Apr;93(4):345-50. doi: 10.1111/aogs.12351. PMID 24575769
- [Background] Hotujec BT, Spencer RJ, Donnelly MJ, Bruggink SM, Rose SL, Al-Niaimi A, Chappell R, Stewart SL, Kushner DM. Transversus abdominis plane block in robotic gynecologic oncology: a randomized, placebo-controlled trial. Gynecol Oncol. 2015 Mar;136(3):460-5. doi: 10.1016/j.ygyno.2014.11.013. Epub 2014 Nov 20. PMID 25462201
- [Background] Torup H, Bogeskov M, Hansen EG, Palle C, Rosenberg J, Mitchell AU, Petersen PL, Mathiesen O, Dahl JB, Moller AM. Transversus abdominis plane (TAP) block after robot-assisted laparoscopic hysterectomy: a randomised clinical trial. Acta Anaesthesiol Scand. 2015 Aug;59(7):928-35. doi: 10.1111/aas.12516. Epub 2015 May 31. PMID 26032118
- [Background] Bharti N, Kumar P, Bala I, Gupta V. The efficacy of a novel approach to transversus abdominis plane block for postoperative analgesia after colorectal surgery. Anesth Analg. 2011 Jun;112(6):1504-8. doi: 10.1213/ANE.0b013e3182159bf8. Epub 2011 Apr 5. PMID 21467560
- [Background] Chetwood A, Agrawal S, Hrouda D, Doyle P. Laparoscopic assisted transversus abdominis plane block: a novel insertion technique during laparoscopic nephrectomy. Anaesthesia. 2011 Apr;66(4):317-8. doi: 10.1111/j.1365-2044.2011.06664.x. No abstract available. PMID 21401554
- [Background] Owen DJ, Harrod I, Ford J, Luckas M, Gudimetla V. The surgical transversus abdominis plane block--a novel approach for performing an established technique. BJOG. 2011 Jan;118(1):24-7. doi: 10.1111/j.1471-0528.2010.02779.x. Epub 2010 Nov 18. PMID 21083866
- [Background] Park SY, Park JS, Choi GS, Kim HJ, Moon S, Yeo J. Comparison of Analgesic Efficacy of Laparoscope-Assisted and Ultrasound-Guided Transversus Abdominis Plane Block after Laparoscopic Colorectal Operation: A Randomized, Single-Blind, Non-Inferiority Trial. J Am Coll Surg. 2017 Sep;225(3):403-410. doi: 10.1016/j.jamcollsurg.2017.05.017. Epub 2017 Jun 10. PMID 28610880
- [Background] Wong DJ, Curran T, Poylin VY, Cataldo TE. Surgeon-delivered laparoscopic transversus abdominis plane blocks are non-inferior to anesthesia-delivered ultrasound-guided transversus abdominis plane blocks: a blinded, randomized non-inferiority trial. Surg Endosc. 2020 Jul;34(7):3011-3019. doi: 10.1007/s00464-019-07097-y. Epub 2019 Sep 4. PMID 31485929
- [Background] Einarsson JI, Sun J, Orav J, Young AE. Local analgesia in laparoscopy: a randomized trial. Obstet Gynecol. 2004 Dec;104(6):1335-9. doi: 10.1097/01.AOG.0000146283.90934.fd. PMID 15572499
- [Background] Tam T, Harkins G, Wegrzyniak L, Ehrgood S, Kunselman A, Davies M. Infiltration of bupivacaine local anesthetic to trocar insertion sites after laparoscopy: a randomized, double-blind, stratified, and controlled trial. J Minim Invasive Gynecol. 2014 Nov-Dec;21(6):1015-21. doi: 10.1016/j.jmig.2014.04.013. Epub 2014 May 2. PMID 24792311
- [Background] Hortu I, Turkay U, Terzi H, Kale A, Yilmaz M, Balci C, Aydin U, Lagana AS. Impact of bupivacaine injection to trocar sites on postoperative pain following laparoscopic hysterectomy: Results from a prospective, multicentre, double-blind randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2020 Sep;252:317-322. doi: 10.1016/j.ejogrb.2020.07.007. Epub 2020 Jul 7. PMID 32653604
- [Background] Barron KI, Lamvu GM, Schmidt RC, Fisk M, Blanton E, Patanwala I. Wound Infiltration With Extended-Release Versus Short-Acting Bupivacaine Before Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2017 Feb;24(2):286-292. doi: 10.1016/j.jmig.2016.11.002. Epub 2016 Nov 14. PMID 27856385